CLINICAL TRIAL: NCT00768365
Title: Cardiovascular Risk in Patients With Non-Functional Adrenal Incidentaloma: Myth or Reality?
Brief Title: Cardiovascular Risk in Patients With Non-Functional Adrenal Incidentaloma
Acronym: adrenal
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: yesim erbil, Istanbul University
Other Study IDs: 2007/675
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-09

CONDITIONS: Adrenal Cortex Neoplasms
Keywords: adrenal incidentaloma; cardiovascular risk
MeSH Terms: conditions — Adrenal Cortex Neoplasms; Adrenal incidentaloma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- group 1: patients with adrenal incidentaloma
- group 2: Thirty-five subjects comparable for sex, age, and BMI were enrolled as a control group (group 2).
- group 3: The other control group (group 3) of 35 healthy individuals matched for sex, age, BMI, metabolic syndrome criteria, cardiovascular risk parameters, menopausal status, smoking status, consumption of alcohol, usage of antihypertensive drugs, insulin or oral hypoglycaemic agents to perform a 1:1 case-control analysis.

SUMMARY:
Between September 2006 and September 2008, 35 patients (32 women and 3 men; mean age 49years with adrenal incidentaloma (AI) were prospectively evaluated at the Department of Endocrinology and General Surgery of Istanbul University, Istanbul Medical Faculty.

All patients with AI underwent physical examination, including waist circumference. Body mass Index (BMI) was calculated as weight (kg)/ height (m) squared. A BMI > 30 was considered an index of obesity. A waist circumference > 88 cm in women and > 95 cm in men was considered the cutoff for visceral obesity in accordance to the Adult Treatment Panel III (ATP III) metabolic syndrome criteria. Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured from the right brachial artery of the patients in a supine position after 10 minutes of rest by using a pneumatic sphygmomanometer by the same doctor.

DETAILED DESCRIPTION:
None of the patients with AI showed specific signs and/or symptoms of hormone excess and none were on hormonal therapy. All patients underwent the following endocrine workup aimed to study the hypothalamic-pituitary-adrenal axis. Serum cortisol, and plasma corticotropin (ACTH) were determined in basal conditions. All patients underwent an overnight 1-mg dexamethasone test. The suppression was adequate when morning cortisol fell below 1.8 lg/dL [21]. If inadequate, a two-day low-dose dexamethasone (DXM) suppression test was performed (2 mg, four times a day for 2 days). Suppressibility was indicated when morning cortisol fell below 1.8 g/dL after the last dose of dexamethasone. In all patients, urinary metanephrine, and normetanephrine excretion were within normal limits and upright plasma aldosterone to plasma renin activity ratio was lower than 20, excluding pheochromocytoma and primary aldosteronism.

Metabolic syndrome criteria Metabolic syndrome criteria were determined according to the ATP III and IDF 2005 guideline and modified as follows; (1) a waist circumference > 88 cm in women and > 94 cm in men, (2) fasting glucose concentrations >100 mg/dl, (3) triglyceride concentrations >150 mg/dl, (4) HDL cholesterol <40 mg/dl in men and <50 mg/dl in women, (5) patients with hypertensive or on antihypertensive medication. Presence of waist criteria plus at least two other criteria were accepted as sufficient for the presence of metabolic syndrome. According to the IDF 2005 guideline, population-specific waist circumferences were also used to evaluate abdominal obesity and metabolic syndrome. For this purpose, a waist circumference of > 83 cm for women and > 95 cm for men were regarded as cut-offs for the presence of abdominal obesity.

Cardiovascular Risk Parameters Cardiovascular Risk Parameters were as follows according to ATP III; (1) family history of premature ischemic heart disease (ischemic heart disease in male first-degree relatives < 55 years, in female first degree relatives < 65 years (2) for male patients age > 45 years, for female patients age > 55 years or being in menopausal state, (3) HDL cholesterol <40 mg/dl in men and <50 mg/dl in women (4) patients with hypertensive or on antihypertensive medication, (5) patients regarded as diabetic (6) current smokers.

ELIGIBILITY:
Inclusion Criteria:

* Between September 2006 and September 2008, 35 patients (32 women and 3 men; mean age 49.1 ± 12 years) with adrenal incidentaloma (AI) were prospectively evaluated at the Department of Endocrinology and General Surgery of Istanbul University, Istanbul Medical Faculty.

Exclusion Criteria:

* Patients with known malignancies and clinical or subclinical hormone secreting tumors were also excluded from this study. Patients with abnormalities of cortisol secretion were also excluded.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study parameters at the patients with AI (group 1) were compared with and control subjects.
  Thirty-five subjects comparable for sex, age, and BMI were enrolled as a control group (group 2). The other control group (group 3) of 35 healthy individuals matched for sex, age, BMI, metabolic syndrome criteria.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Doppler ultrasonography | at the time of the detection of the adrenal incidentaloma

CONTACTS AND LOCATIONS:
Overall Officials: yesim erbil, prof, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Capa, Turkey (Türkiye)

REFERENCES:
- [Background] Ermetici F, Malavazos AE, Corbetta S, Morricone L, Dall'Asta C, Corsi MM, Ambrosi B. Adipokine levels and cardiovascular risk in patients with adrenal incidentaloma. Metabolism. 2007 May;56(5):686-92. doi: 10.1016/j.metabol.2006.12.018. PMID 17445545
- [Derived] Erbil Y, Ozbey N, Barbaros U, Unalp HR, Salmaslioglu A, Ozarmagan S. Cardiovascular risk in patients with nonfunctional adrenal incidentaloma: myth or reality? World J Surg. 2009 Oct;33(10):2099-105. doi: 10.1007/s00268-009-0178-0. PMID 19649755